CLINICAL TRIAL: NCT07121790
Title: The Use of Magnesium (Mg)-Based Absorbable DrillPins in Hammertoe Deformity Correction: a Feasibility Study
Brief Title: Mg Alloy DrillPins in Hammertoe Deformity Correction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bioretec Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 243-03-CI-01
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Hammertoe; Hammer Toe Syndrome
Keywords: deformity; device; Hammertoe surgery; absorbable implant; osteotomy fixation; DrillPin; RemeOs
MeSH Terms: conditions — Hammer Toe Syndrome; Congenital Abnormalities

STUDY DESIGN:
Intervention Model Description: Single-arm interventional study in which all enrolled participants receive the investigational device, the RemeOs™ DrillPin, for surgical correction of hammertoe deformities. All patients are followed using a standardized clinical and radiographic assessment schedule.
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hammertoe correction surgery with Mg-based DrillPins (Experimental)
  Interventions: Device: Implant Mg-based RemeOs™ drillpins

INTERVENTIONS:
Device: Implant Mg-based RemeOs™ drillpins — This is a first-in-human clinical feasibility study of a novel absorbable magnesium-zinc-calcium alloy DrillPin (RemeOs™) for internal fixation during surgical correction of hammertoe deformities in adult patients. The implant is investigational, not CE-marked, and represents an alternative to conventional stainless steel or titanium K-wires commonly used in toe correction surgery.
  The RemeOs™ DrillPin is designed to provide mechanical stability during osteotomy healing and gradually resorbs over 2-3 years, potentially eliminating the need for secondary implant removal.
  The study focuses on evaluating safety, performance, and implant resorption using standardized clinical and radiographic assessments. The DrillPin is made from the same magnesium alloy (ZX00) as the CE-marked RemeOs™ Screw, which has demonstrated clinical safety and performance in prior applications.

SUMMARY:
This is a prospective, single-arm clinical feasibility study evaluating the safe application of a novel lean absorbable magnesium-zinc-calcium alloy (ZX00) drill pin (RemeOs™ DrillPin) for the surgical correction of hammertoe deformities. A total of 20 adult patients will be enrolled. All participants will receive the investigational implant without a comparator or control group. The study focuses on feasibility, safety, and functional outcomes following implantation.

DETAILED DESCRIPTION:
This single-arm, open-label, monocenter clinical investigation is conducted in accordance with ISO 14155 to evaluate the safety and performance of the RemeOs™ DrillPin, an absorbable magnesium-zinc-calcium alloy (ZX00) implant, for internal fixation during hammertoe correction surgery in adult patients.

Eligible participants are adults aged 18 years and older with hammertoe deformity of the lesser toes requiring surgical correction, with or without concomitant hallux valgus surgery. The RemeOs™ DrillPin is designed to provide mechanical stability during osteotomy healing and gradually resorbs over time, potentially eliminating the need for implant removal and reducing infection risk through primary wound closure.

Primary objectives include assessing implantation success-defined as low pain levels (VAS <3) and good or fair toe alignment according to the AOFAS Lesser Metatarsophalangeal-Interphalangeal Scale (AOFAS-LMIS)-at 12 weeks postoperatively, as well as short-term safety, measured by the incidence of adverse and serious adverse device events (ADEs/SADEs).

Secondary assessments include clinical evaluation of pain, wound healing, DIP joint function, and neurovascular status at 2, 4, 6, and 12 weeks, and at 12 and 36 months. Radiographic assessments will monitor alignment, gas formation, and osteolysis at each follow-up, with CT imaging at 12 and 36 months to evaluate implant resorption and potential local effects.

This feasibility study aims to generate initial clinical data on the use of absorbable magnesium-based implants in forefoot surgery and to assess their potential to maintain deformity correction without the need for implant retrieval.

ELIGIBILITY:
Inclusion Criteria:

* Hammertoe deformity of the lesser toes, with or without accompanying surgery of a hallux valgus deformity
* Written informed consent of the participant
* Female and male patients aged 18 years and more
* Subject has been informed of the nature of the study, agrees to participate and signs the approved consent form
* Subject is able and willing to comply with all assessments in the study.
* Female patients in childbearing age perform a pregnancy test prior to inclusion

Exclusion Criteria:

* Pathological bone lesions (e.g., bone cysts or osteomyelitis)
* Underlying diseases (kidney diseases, diabetes mellitus)
* Chronic alcoholics
* Severe mental illness
* Pregnant or breastfeeding women
* Inability or unwillingness to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with pain score <3 on the Visual Analogue Scale (VAS) (criterion of successful implantation) | At 12 weeks postoperatively
  This outcome is one of two predefined criteria used to determine successful implantation. Pain will be measured using the Visual Analogue Scale (VAS), ranging from 0 (no pain) to 10 (worst pain). A score of less than 3 at 12 weeks postoperatively is considered a successful pain outcome
Number of participants with good or fair alignment on the AOFAS Lesser Metatarsophalangeal-Interphalangeal Scale (AOFAS-LMIS) (criterion of successful implantation) | At 12 weeks postoperatively
  This is one of two predefined criteria for successful implantation. Toe alignment will be assessed at 12 weeks postoperatively using the alignment domain of the AOFAS-LMIS. In this subscale, alignment is scored as follows:
  15 points: Good alignment (toe well aligned) 8 points: Fair alignment (some malalignment without symptoms) 0 points: Poor alignment (obvious symptomatic malalignment)
  An alignment score of 8 or 15 points is considered a successful outcome.
Number of participants with at least one adverse device event (ADE) or serious adverse device event (SADE) | From surgery to 12 weeks postoperatively
  This outcome measures the short-term safety of the investigational device. Safety will be assessed by recording the occurrence, type, severity, and investigator-assessed relationship of all adverse device events (ADEs) and serious adverse device events (SADEs) from surgery through 12 weeks postoperatively. Data will be collected through clinical evaluations, subject interviews, and medical record review.

SECONDARY OUTCOMES:
Degree of DrillPin resorption | 12 and 36 months postoperatively
  The extent of implant resorption will be assessed using CT (computed tomography) imaging at 12 and 36 months postoperatively. Resorption will be classified as one of the following categories:
  * Not visible/slight
  * Partial (25-75%)
  * Complete (implant not visible)
  Each participant will be assigned to one resorption category based on imaging findings.
Number of participants with radiographic evidence of subcutaneous gas formation | 12 and 36 months postoperatively
  Presence or absence of subcutaneous gas cavities will be assessed using CT imaging at 12 and 36 months postoperatively.
  A binary Yes/No result will be recorded per participant.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Holweg, Prof. Dr., Principal Investigator — Department of Orthopaedics and Trauma, Medical University of Graz

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. The study data are pseudonymized and retained only by the investigator site with no access to direct identifiers by the sponsor. The sponsor only receives pseudonymized data for analysis and regulatory use.

REFERENCES:
- [Result] Klammer G, Baumann G, Moor BK, Farshad M, Espinosa N. Early complications and recurrence rates after Kirschner wire transfixion in lesser toe surgery: a prospective randomized study. Foot Ankle Int. 2012 Feb;33(2):105-12. doi: 10.3113/FAI.2012.0105. PMID 22381341
- [Result] Holweg P, Berger L, Cihova M, Donohue N, Clement B, Schwarze U, Sommer NG, Hohenberger G, van den Beucken JJJP, Seibert F, Leithner A, Loffler JF, Weinberg AM. A lean magnesium-zinc-calcium alloy ZX00 used for bone fracture stabilization in a large growing-animal model. Acta Biomater. 2020 Sep 1;113:646-659. doi: 10.1016/j.actbio.2020.06.013. Epub 2020 Jun 14. PMID 32553919
- [Result] Bostman O, Pihlajamaki H. Routine implant removal after fracture surgery: a potentially reducible consumer of hospital resources in trauma units. J Trauma. 1996 Nov;41(5):846-9. doi: 10.1097/00005373-199611000-00013. PMID 8913214